CLINICAL TRIAL: NCT01343290
Title: A Single-Dose, Open-Label, Randomized, 2-Period, 2-Sequence, Crossover Study to Determine the Effect of Food Coadministration on the Pharmacokinetics of 300 mg Canagliflozin in Healthy Subjects
Brief Title: The Effect of Food on the Administration of Canagliflozin in Healthy Adult Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Johnson & Johnson Pharmaceutical Research & Development, L.L.C. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: CR018016; 284317541043
Record Dates: First submitted 2011-04-01; First posted 2011-04-28 (Estimated); Last update posted 2012-10-02 (Estimated); Status verified 2012-09

CONDITIONS: Healthy
Keywords: Canagliflozin (JNJ-28431754); Pharmacokinetic; Oral Bioavailability; Food effect
MeSH Terms: interventions — Canagliflozin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 001 (Experimental): Canagliflozin Type = 1 unit = mg number = 300 form = tablet route = oral use. Single tablet taken with or without a meal during 2 treatment periods
  Interventions: Drug: Canagliflozin

INTERVENTIONS:
Drug: Canagliflozin — Type = 1, unit = mg, number = 300, form = tablet, route = oral use. Single tablet taken with or without a meal during 2 treatment periods

SUMMARY:
The purpose of this study is to assess the effect of food on the absorption of canagliflozin in the body when canagliflozin is taken with and without food by healthy volunteers

DETAILED DESCRIPTION:
This is a single-center, single-dose, open-label (volunteers will know the identity of assigned treatment), randomized (one of 2 study drug sequences assigned by chance) study to evaluate the oral bioavailability (the degree to which the drug is absorbed in the body when taken orally by mouth) of canagliflozin when taken with and without food in healthy volunteers. Healthy Volunteers will take 1 canagliflozin tablet orally for 1 day in 2 treatment periods (canagliflozin will be taken with food in 1 treatment period and canagliflozin will be taken without food in 1 treatment period); the 2 treatment periods will be separated by a 10- to 14-day washout period.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers with a body mass index between 18 and 30 kg/m2 (inclusive) and body weight not less than 50 kg

Exclusion Criteria:

* of or current medical illness deemed clinically significant by the Investigator (study physician)

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2011-04; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Concentration of canagliflozin in plasma samples | For up to 8 days

SECONDARY OUTCOMES:
Adverse events reported | Up to approximately 34 days
Vital signs measurements | Up to approximately 34 days
Results from clinical chemistries performed | Up to approximately 34 days
Results from 12-lead ECGs performed | Up to approximately 34 days

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson Pharmaceutical Research & Development, L.L. C. Clinical Trial, Study Director — Johnson & Johnson Pharmaceutical Research & Development, L.L.C.

REFERENCES:
- [Derived] Devineni D, Manitpisitkul P, Murphy J, Stieltjes H, Ariyawansa J, Di Prospero NA, Rothenberg P. Effect of food on the pharmacokinetics of canagliflozin, a sodium glucose co-transporter 2 inhibitor, and assessment of dose proportionality in healthy participants. Clin Pharmacol Drug Dev. 2015 Jul;4(4):279-86. doi: 10.1002/cpdd.151. Epub 2014 Dec 11. PMID 27136908